CLINICAL TRIAL: NCT05779774
Title: WayToServe Plus: In-service Professional Development Component to Improve Responsible Alcohol Service Ph II
Brief Title: WayToServePlus: Improving Responsible Alcohol Service Ph II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Pacific Institute for Research and Evaluation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 0338; 4R44AA029364-02 (NIH)
Record Dates: First submitted 2023-02-07; First posted 2023-03-22 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking; Alcohol Intoxication; Alcohol Use, Unspecified
Keywords: Alcohol service; Driving under influence; DWI prevention; Safe alcohol service
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication; Driving Under the Influence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Premises are unaware of the pseudo patrons sent in for data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WayToServe Plus In-service Component (Experimental): Intervention group of servers to participate in Facebook group.
  Interventions: Behavioral: WayToServe Plus In-service Component
- WayToServe Training Only (Experimental): Control group of servers who do not participate in Facebook group and receive WayToServe Training only.
  Interventions: Behavioral: WayToServe Training Only

INTERVENTIONS:
Behavioral: WayToServe Plus In-service Component — Investigators will test WayToServe Plus in-service component's ability to increase refusal of service to intoxicated patrons in a randomized trial. A two-group randomized field trial (WayToServe training only [comparison control] v. WayToServe training plus WayToServe Plus in-service component [intervention]) with 2 assessment rounds (Baseline, Posttest) will yield a 2 factorial design. Investigators will randomly assign premises to WayToServe training and WayToServe Plus after baseline in Month 18, stratified by state and location. Remaining premises will receive WayToServe Training Only. All premises will be recruited to have servers complete WayToServe training. Servers in intervention group will be accepted into a Facebook private group after WayToServe training to receive in-service component with ~3 posts per week for 12 months. In Months 30-32, all premises will be posttested with PiP assessments (blind to condition).
  Arms: WayToServe Plus In-service Component
Behavioral: WayToServe Training Only — Investigators will test WayToServe Plus in-service component's ability to increase refusal of service to intoxicated patrons in a randomized trial. A two-group randomized field trial (WayToServe Training Only [comparison control] v. WayToServe Plus In-service Component [intervention]) with 2 assessment rounds (Baseline, Posttest) will yield a 2 factorial design. Investigators will randomly assign premises to WayToServe Traiing Only after baseline in Month 18, stratified by state and location. In Months 30-32, all premises will be posttested with PiP assessments (blind to condition).
  Arms: WayToServe Training Only

SUMMARY:
Responsible beverage service (RBS) training for alcohol servers is a promising intervention for reducing driving while intoxicated (DWI) by alcohol. Training, certification, and in-service contact improves professionalism and effectiveness of prevention interventions delivered by community members such as alcohol servers. This SBIR Fast-track project will develop and test an in-service professional development component to the WayToServe® online RBS training to improve the effectiveness of RBS training in order to make further gains in reducing problem alcohol behavior in communities.

DETAILED DESCRIPTION:
Among the interventions targeting driving while intoxicated (DWI) by alcohol, Responsible Beverage Service (RBS) training of alcohol servers has shown promise. RBS training is currently required or incentivized by 36 U.S. states and California will require it starting in 2022. The research team has shown that an online RBS training, named WayToServe®, was effective in two randomized trials. These results filled a gap in the literature on RBS training that is limited by the lack of randomized trials, poor measurement of training implementation, and almost exclusive focus on live training when online training predominates. The goal of this SBIR Fast-track research is to develop and test an in-service professional development component for alcohol servers trained by WayToServe to improve its effectiveness. It is intended to motivate servers to implement the RBS skills in the face of common barriers, provide support for RBS actions from a "community" of alcohol servers, and prevent natural degradation of skills over time. Rationale for this product is provided by past research showing that training, certification, and in-service contact improves professionalism and efficacy of community prevention interventions. Scientific premise is provided by the positive results of our trials on the WayToServe® training. The in-service component will be delivered through the WayToServe Facebook page that currently is "followed" by over 20,000 alcohol servers trained by WayToServe. The specific aims of Phase I are to: 1) develop content of in-service professional development on RBS skills with a) premises owners/ managers interviews and b) alcohol servers in New Mexico and Washington State trained by the WayToServe online RBS training through focus group discussions; 2) produce a prototype WayToServe Plus in-service professional development component in flowcharts and an initial library of Facebook posts, including text, graphics, and interactive elements and evaluate it for acceptability, usability, and engagement in focus groups and field pilot trial with alcohol servers in New Mexico and Washington State trained by the WayToServe online RBS training, and 3) determine feasibility of WayToServe Plus in-service professional development component and develop evaluation plans for Phase II research. Milestones will be an EAB-approved Phase I research plans and development of the content outline and WayToServe Plus prototype, evaluation of WayToServe Plus prototype, and feasibility assessment of the WayToServe Plus in-service professional development component. Phase II specific aims will achieve the milestones of full production of WayToServe Plus and a randomized trial testing its effectiveness by: 4) producing the full WayToServe Plus in-service professional development component and 5) conducting a randomized trial with 160 alcohol premises in New Mexico and Washington State evaluating effectiveness of WayToServe Plus on refusal of sales to PiP (primary outcome). The SBIR research is innovative as WayToServe Plus will be the first continuous in-service professional development for RBS and will increase the WayToServe training's effectiveness and commercial advantage with alcohol servers and corporate clients.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Own/manage a licensed premises or be an alcohol server (waitress, waiter or bartender)
* Have completed the WayToServe responsible beverage service training (Phase I only)
* Be proficient in English
* Consent to participate

Exclusion Criteria:

* Have a family/household member already participating in project • Younger than 19 years old (18 and younger cannot legally serve alcohol in either state)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1172 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Refusal rate of alcohol service to apparently-intoxicated patrons | Change in refusal rate between baseline and 1 year posttest assessments
  Primary outcome measure, refusal rate of alcohol service to apparently-intoxicated patrons, will be obtained via a pseudo-intoxicated patron (PiP) assessment. Confederate buyers will feign intoxication and record if servers agree to serve them an alcoholic beverage. PiP protocol presents a server with the most overt situation in which alcohol service should be refused, (i.e., when a patron is showing clear signs of intoxication), models behavior of patrons most at risk, and is relatively low cost.

CONTACTS AND LOCATIONS:
Overall Officials: David Buller, PhD, Principal Investigator — Klein Buendel, Inc.; Gill Woodall, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (1):
- Klein Buendel, Inc, Golden, Colorado, United States

REFERENCES:
- [Derived] Woodall WG, Buller D, Saltz R, Martinez L. Professional Development to Improve Responsible Beverage Service Training: Formative Research Results and Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Jan 24;13:e49680. doi: 10.2196/49680. PMID 38265847

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT05779774/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT05779774/ICF_001.pdf